CLINICAL TRIAL: NCT03909750
Title: Use of Autologous Stem/Stromal Cells in Chronic Lung Disorders: Obstructive (COPD) and Restrictive (RLD)
Brief Title: Use of Autologous Stem/Stromal Cells In Chronic Lung Disorders: Obstructive (COPD) & Restrictive (RLD)
Acronym: cSVF-Lung
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn [COVID restrictions prevent patient enrollment or treatment. Clinical Trial facility is being closed due to viral limitations and loss of staff to perform]
Sponsor: Healeon Medical Inc (Industry)
Collaborators: Robert W. Alexander, MD (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GARM 2 Lung
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: COPD; Respiratory Insufficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lipoaspiration Microcannula ARM 1 (Experimental): Acquisition of Adipose-Derived tissue Stromal Vascular Fraction (AD-tSVF) via closed syringe harvest subdermal fat
  Interventions: Procedure: Lipoaspiration
- Isolation-Concentration Adipose cSVF ARM 2 (Experimental): Isolation of cellular stem/stromal cells from subdermal adipose-derived cellular stromal vascular fraction (AD-cSVF)
  Interventions: Procedure: AD-cSVF
- Normal Saline IV ARM 3 (Experimental): Sterile Normal Saline IV with cSVF
  Interventions: Procedure: Normal Saline IV

INTERVENTIONS:
Procedure: Lipoaspiration — Close syringe microcannula harvesting subdermal fat and perivascular stem/stromal cells
  Arms: Lipoaspiration Microcannula ARM 1
Procedure: AD-cSVF — Isolation of AD-cSVF
  Arms: Isolation-Concentration Adipose cSVF ARM 2
Procedure: Normal Saline IV — Normal Saline IV containing AD-cSVF
  Arms: Normal Saline IV ARM 3

SUMMARY:
Pulmonary Disorders are often categorized as Obstructive or Restrictive disorders. This study will establish two channels of investigation, one group within each type of pulmonary dysfunction. State-of-the-Art Objective analytics will be employed to track patients from baseline and 6 month intervals for up to one year.

Chronic Obstructive Pulmonary Disease (COPD) is a lung-related disorder that is characterized by long-term, often progressive state of poor airflow. Primary symptoms include low oxygen tension, shortness of breath, productive cough, and broncho-pulmonary inflammation and interference with oxygen-carbon dioxide exchange. COPD is generally considered those who are able to better inspire air than to expel. Restrictive lung dysfunctions are generally considered those who are unable to achieve full inspiration function. Both can create some of the same symptoms, low Oxygen exchange, activity intolerance of exertion, shortness of breath (SOB), Pulmonary Hypertension, Loss of lung structure, Pneumothorax (in emphysema), may mandate supplemental Oxygen therapy, failure of airway mucus management (chronic bronchitis, bronchiectasis, etc), and other failure of lung function issues.

Restrictive lung disorders represent a group of pulmonary function losses which are due to acquired fibrosis, congenital fibrotic disorders, functional airway damage (scarring), vascular abnormalities in arterial/venous supply,

Air pollution and tobacco smoking, chemical inhalation damage, etc. are felt to be common contributor of these issues. Diagnostic testing is based on poor airflow measured by lung function studies and whose symptoms do not improve much with anti-asthma bronchodilators, steroids, and a variety of combination of topical medications.

Study is an interventional study to document the safety and efficacy of use of cSVF in chronic broncho-pulmonary disease within both groups.

DETAILED DESCRIPTION:
Pulmonary Disorders, including both COPD & Restrictive Lung Disease (RLD) are often treated by limiting exposure to poor air quality, but there is no cure at this time. Most commonly, the patients are treated upon exacerbations, usually with some combination of inhalers, steroids, and medications which have proven to be ineffective other than addressing symptoms and trying to return to baseline symptom help. In addition, many attempted efforts are aimed at environmental changes, therapy include smoking cessation, vaccinations, respiratory rehabilitation, and attempts of use of bronchodilators and topical and systemic steroids. Many must resort to supplemental oxygen therapy, lung transplantation, and antibiotic supportive therapy during exacerbations.

As of 2013, COPD involve approximately 5% of the global populations (approximately 330 million). Most commonly it occurs approximately equally between men/women and result in about 3 million deaths per year. Estimates of economic costs are estimated to be more than 2.1 trillion dollars in 2010.

This study includes microcannula harvesting of subdermal adipose tissues, incubation, digestion and isolation of AD-cSVF. This stromal cellular pellet (without actual extracellular matrix or stromal elements) is then suspended in 500 cc sterile Normal Saline (NS) and deployed via peripheral intravenous route. Evaluations of safety issues are measured at intervals (both severe and non-severe categories) and by repeated pulmonary function studies.

Most pulmonary function tests are, at best some help, but there is now a remarkable testing that is substantially more informative than standard flow measurements, as they include extensive anatomical and functional insights using High Resolution Computerized Tomography (HRCT) Lung. This protocol allows for direct evidence of the air trapping, lung volume capabilities, and three dimensional imaging of the airways and lungs themselves. This modality will be the primary comparative between baseline and 6 month post-therapy in determination of the status and changes than can be demonstrated following use of cellular stromal vascular fraction (cSVF). After isolation and concentration of the stem/stromal cells via digestive processing, deployment of such cellular elements are believed to engraft within the lung capillary tissues. Engraftment is not currently believed to be the primary elements following parenteral (IV) placement. Rather, it is believed to represent the paracrine secretory and communication between cell-to-cell or cell-to-matrix which communicates via exosomal and microvesicular contents that are released to influence the local niche (microenvironment). Via transfer of microRNA (mRNA) or mitoRNA (miRNA), stem cells are able to help other pulmonary cells replace or repair damaged elements associated with lung disorders. Further, these secretions and growth factor/cytokines availability have a positive influence on the small capillaries within the lung parenchyma, thereby likely to improve the gas exchange function within the lungs.

Tracking of oxygen saturation (at rest and activity), use of inhalers or other rescue effort reduction, reduction of oxygen supplement, and improved respiratory efforts will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Documented COPD or RLD by qualified Medical Provider
* History of Pulmonary Function Deficits or supplemental oxygen therapy

Exclusion Criteria:

* Cancer of the Lung
* Patient's on chemotherapy or radiation for Cancer (or History within 5 years)
* Inability to comply with Baseline and 6 month post-treatment HDCT lungs
* General health or inability or unwillingness or ability to provide informed consent for study
* History of lung transplantation
* Life expectancy of <3 months due to concomitant illnesses
* Exposure to any investigational drug of procedure within 1 month prior to study enrollment which may interfere with interpretation of outcomes
* Illness which, in investigator's judgement, may interfere with patient's ability of comply with protocol, compromise patient safety, ability to provide informed consent or interfere with the interpretation of study outcomes.
* Subjects with chronic immunosuppressive or chemotherapeutic medication.
* Known drug or alcohol dependence or other factors which may interfere with study conduct or interpretation of result in opinion of investigators.
* Subjects with documented Alpha 2 Antitrypsin Deficiency (inherited lung and liver disorder)
* Patient with history of Hepatitis (except Hepatitis A history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety-Pulmonary Function: occurrence or frequency of adverse or severe adverse events during study | 6 months evaluate function and adverse events
  Pulmonary Function as occurrence or frequency of adverse or severe adverse events during study

SECONDARY OUTCOMES:
High Resolution Computerized Tomography - Lungs Fluidda Analysis | Baseline and 6 month Comparative Study
  Fluidda Pulmonary Objective Analytics

CONTACTS AND LOCATIONS:
Overall Officials: Glenn C Terry, MD, Principal Investigator — Global Alliance for Regenerative Medicine (GARM-HN)
Locations (2):
- Global Alliance for Regenerative Medicine-USA, Stevensville, Montana, United States
- Global Alliance of Regenerative Medicine (GARM) International, Roatán, Hn, Honduras

REFERENCES:
- [Result] Decramer M, Janssens W, Miravitlles M. Chronic obstructive pulmonary disease. Lancet. 2012 Apr 7;379(9823):1341-51. doi: 10.1016/S0140-6736(11)60968-9. Epub 2012 Feb 6. PMID 22314182
- [Result] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Result] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Result] Mahler DA. Mechanisms and measurement of dyspnea in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2006 May;3(3):234-8. doi: 10.1513/pats.200509-103SF. PMID 16636091
- [Result] Holland AE, Hill CJ, Jones AY, McDonald CF. Breathing exercises for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD008250. doi: 10.1002/14651858.CD008250.pub2. PMID 23076942
- [Result] Kennedy SM, Chambers R, Du W, Dimich-Ward H. Environmental and occupational exposures: do they affect chronic obstructive pulmonary disease differently in women and men? Proc Am Thorac Soc. 2007 Dec;4(8):692-4. doi: 10.1513/pats.200707-094SD. PMID 18073405
- [Result] Devereux G. ABC of chronic obstructive pulmonary disease. Definition, epidemiology, and risk factors. BMJ. 2006 May 13;332(7550):1142-4. doi: 10.1136/bmj.332.7550.1142. No abstract available. PMID 16690673
- [Result] Foreman MG, Campos M, Celedon JC. Genes and chronic obstructive pulmonary disease. Med Clin North Am. 2012 Jul;96(4):699-711. doi: 10.1016/j.mcna.2012.02.006. Epub 2012 Mar 6. PMID 22793939
- [Result] O'Donnell DE. Hyperinflation, dyspnea, and exercise intolerance in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2006 Apr;3(2):180-4. doi: 10.1513/pats.200508-093DO. PMID 16565429
- [Result] Mackay AJ, Hurst JR. COPD exacerbations: causes, prevention, and treatment. Med Clin North Am. 2012 Jul;96(4):789-809. doi: 10.1016/j.mcna.2012.02.008. Epub 2012 Mar 16. PMID 22793945
- [Result] Puhan MA, Gimeno-Santos E, Scharplatz M, Troosters T, Walters EH, Steurer J. Pulmonary rehabilitation following exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD005305. doi: 10.1002/14651858.CD005305.pub3. PMID 21975749
- [Result] Saxena A, Watkin SW. Bilateral malignant testicular carcinoid. Br J Urol. 1990 Mar;65(3):302-3. doi: 10.1111/j.1464-410x.1990.tb14738.x. No abstract available. PMID 2337756
- [Result] Kew KM, Seniukovich A. Inhaled steroids and risk of pneumonia for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2014 Mar 10;2014(3):CD010115. doi: 10.1002/14651858.CD010115.pub2. PMID 24615270
- [Result] COPD Working Group. Long-term oxygen therapy for patients with chronic obstructive pulmonary disease (COPD): an evidence-based analysis. Ont Health Technol Assess Ser. 2012;12(7):1-64. Epub 2012 Mar 1. PMID 23074435
- [Result] Bradley JM, O'Neill B. Short-term ambulatory oxygen for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD004356. doi: 10.1002/14651858.CD004356.pub3. PMID 16235359
- [Result] Vollenweider DJ, Jarrett H, Steurer-Stey CA, Garcia-Aymerich J, Puhan MA. Antibiotics for exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Dec 12;12:CD010257. doi: 10.1002/14651858.CD010257. PMID 23235687
- [Result] Inamdar AC, Inamdar AA. Mesenchymal stem cell therapy in lung disorders: pathogenesis of lung diseases and mechanism of action of mesenchymal stem cell. Exp Lung Res. 2013 Oct;39(8):315-27. doi: 10.3109/01902148.2013.816803. Epub 2013 Aug 30. PMID 23992090
- [Result] Conese M, Piro D, Carbone A, Castellani S, Di Gioia S. Hematopoietic and mesenchymal stem cells for the treatment of chronic respiratory diseases: role of plasticity and heterogeneity. ScientificWorldJournal. 2014 Jan 19;2014:859817. doi: 10.1155/2014/859817. eCollection 2014. PMID 24563632
- [Result] McQualter JL, Anthony D, Bozinovski S, Prele CM, Laurent GJ. Harnessing the potential of lung stem cells for regenerative medicine. Int J Biochem Cell Biol. 2014 Nov;56:82-91. doi: 10.1016/j.biocel.2014.10.012. Epub 2014 Oct 15. PMID 25450456
- [Result] Tzouvelekis A, Ntolios P, Bouros D. Stem cell treatment for chronic lung diseases. Respiration. 2013;85(3):179-92. doi: 10.1159/000346525. Epub 2013 Jan 29. PMID 23364286
- [Result] Tzouvelekis A, Laurent G, Bouros D. Stem cell therapy in chronic obstructive pulmonary disease. Seeking the Prometheus effect. Curr Drug Targets. 2013 Feb;14(2):246-52. doi: 10.2174/1389450111314020009. PMID 23256721